CLINICAL TRIAL: NCT01737827
Title: A Phase II, Open Label, Single Arm, Multicenter Study of INC280 Administered Orally in Adults With Advanced Hepatocellular Carcinoma
Brief Title: Study Efficacy and Safety of INC280 in Patients With Advanced Hepatocellular Carcinoma.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study recruitment was ended due to difficulties in identifying subjects who meet the eligibility criteria and therefore the study never reached its planned sample size per protocol. The study termination was not due to any safety concerns.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CINC280X2201
Record Dates: First submitted 2012-11-12; First posted 2012-11-30 (Estimated); Results first posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Advanced Hepatocellular Carcinoma With c-MET Dysregulation
Keywords: INC280; capmatinib; advanced hepatocellular carcinoma; c-MET pathway dysregulation
MeSH Terms: interventions — capmatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- INC280 (Experimental): The protocol consisted of two independent parts (Dose-Determining Part and Dose Expansion Part). Patients were treated with INC280 300 mg twice a day in the Dose-Determining Part. The dose for the Expansion Part could be lower, equal or higher than in the Dose-Determining Part and was determined after the Dose Determining Part at the dose decision analysis.
  Interventions: Drug: INC280

INTERVENTIONS:
Drug: INC280 — INC280 was administered orally on a continuous twice a day (BID) dosing schedule, from Day 1 until Day 21 of each 21-day cycle. INC280 was initially supplied as hard gelatin capsules and subsequently also as film-coated tablets.
  Other Names: capmatinib

SUMMARY:
This study is to find out if INC280 is safe and has beneficial effects in patients with advanced hepatocellular carcinoma known to have dysregulation of c-MET pathway.

DETAILED DESCRIPTION:
This study was designed as a Phase II, single arm, open-label, multicenter study to evaluate the safety and efficacy of INC280 as first-line treatment in patients with advanced hepatocellular carcinoma (HCC) who were not eligible for or had disease progression after surgical or locoregional therapies, with c-MET dysregulation.

The study included a Dose-Determining Part and a Dose Expansion Part. Pharmacokinetic and safety profiles of INC280 in the setting of liver dysfunction were determined in the Dose-Determining Part. The Dose Expansion Part started when the appropriate dose for patients with liver dysfunction was determined based on pharmacokinetics (PK) and safety data from the Dose-Determining Part and other INC280 clinical studies. The initial dose of INC280 assessed during the dose expansion part was 600 mg twice daily (BID) administered as capsules of 50 mg. Later during the dose expansion part, a tablet with higher dosage strengths (50 mg, 150 mg, and 200 mg) was developed and introduced to improve the convenience of study drug administration for patients. PK data on INC280 tablet at 400 mg BID from other studies (NCT01324479, NCT01546428 and NCT01610336) showed that systemic exposure to INC280 was in the range of that achieved with the capsule at 600 mg BID.

During the Dose Expansion part of the study, Novartis halted the enrollment in Dec-2016 due to difficulty in identifying patients who met the definition of c-MET high as defined in the inclusion criteria. Patients who were already enrolled and signed the informed consent were allowed to continue in the study according to the protocol. The enrollment halt was not a consequence of any safety concerns.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed c-MET pathway dysregulation.
* Advanced hepatocellular carcinoma which could not be suitable for treatment with locoregional therapies or has progressed following locoregional therapy.
* Measurable disease as determined by RECIST version 1.1.
* Current cirrhotic status of Child-Pugh class A with no encephalopathy.
* Eastern Cooperative Oncology Group (ECOG) performance status < or = 2.

Exclusion Criteria:

* Received any prior systemic chemotherapy or molecular-targeted therapy for hepatocellular carcinoma such as sorafenib.
* Previous treatment with c-MET inhibitor or hepatocyte growth factor targeting therapy.
* Previous local therapy completed less than 4 weeks prior to dosing and, if present, any acute toxicity > grade 1.
* Known active bleeding (e.g. bleeding from gastro-intestinal ulcers or esophageal varices) within 2 months prior to screening or with history or evidence of inherited bleeding diathesis or coagulopathy.
* Clinically significant venous or arterial thrombotic disease within past 6 months.
* History of acute or chronic pancreatitis, surgery of pancreas or any risk factors that may increase risk of pancreatitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-03-25 (Actual); Primary Completion 2023-04-24 (Actual); Study Completion 2023-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- China (3):
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Xi’an, Shanxi
  - Novartis Investigative Site, Hangzhou, Zhejiang
- Novartis Investigative Site, Hong Kong, Hong Kong
- Novartis Investigative Site, Singapore, Singapore
- Thailand (2):
  - Novartis Investigative Site, Khon Kaen, THA
  - Novartis Investigative Site, Bangkok

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

REFERENCES:
- [Derived] Qin S, Chan SL, Sukeepaisarnjaroen W, Han G, Choo SP, Sriuranpong V, Pan H, Yau T, Guo Y, Chen M, Ren Z, Xu J, Yen CJ, Lin ZZ, Manenti L, Gu Y, Sun Y, Tiedt R, Hao L, Song W, Tanwandee T. A phase II study of the efficacy and safety of the MET inhibitor capmatinib (INC280) in patients with advanced hepatocellular carcinoma. Ther Adv Med Oncol. 2019 Dec 11;11:1758835919889001. doi: 10.1177/1758835919889001. eCollection 2019. PMID 31853265

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 9 investigative sites in 4 countries.
Pre-assignment Details: Evidence of c-MET pathway dysregulation had to be available to be eligible to participate in this study.
  After the molecular pre-screening, screening assessments had to be done within 14 days prior to the first dose of INC280.
  The study included a Dose-Determining Part designed to identify an appropriate dose for patients with hepatocellular carcinoma (HCC) and a Dose Expansion part designed to estimate the efficacy in patients with HCC with different levels of c-MET expression.
Groups:
- CINC280 300 mg BID Capsule: INC280 300 mg orally twice daily (BID) as capsule
- CINC280 600 mg BID Capsule: INC280 600 mg orally twice daily (BID) as capsule
- CINC280 400 mg BID Tablet: INC280 400 mg orally twice daily (BID) as tablet
Period: Overall Study
Arm/Group | CINC280 300 mg BID Capsule | CINC280 600 mg BID Capsule | CINC280 400 mg BID Tablet
Started (All patients enrolled) | 8 | 28 | 2
Dose-Determining Part (Patients enrolled in the Dose-Determining part of the study) | 8 | 0 | 0
Dose Expansion Part: c-MET High (Patients enrolled in the Dose Expansion part of the study with c-MET High) | 0 | 8 | 2
Dose Expansion Part: c-MET Low (Patients enrolled in the Dose Expansion part of the study with c-MET Low) | 0 | 20 | 0
Safety Set (All patients who received at least one dose of INC280. Patients were analyzed according to the treatment they actually received.) | 9 | 27 | 2
Completed | 0 | 0 | 0
Not Completed | 8 | 28 | 2
Not completed — Adverse Event | 3 | 6 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Physician Decision | 0 | 2 | 0
Not completed — Progressive Disease | 5 | 16 | 2
Not completed — Study Terminated by Sponsor | 0 | 1 | 0
Not completed — Subject/Guardian Decision | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CINC280 300 mg BID Capsule | CINC280 600 mg BID Capsule | CINC280 400 mg BID Tablet | Total
Number analyzed (Participants) | 8 | 28 | 2 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (7.97) | 55.0 (9.34) | 53.5 (0.71) | 55.6 (8.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 0 | 4
  Male | 7 | 25 | 2 | 34
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 8 | 28 | 2 | 38
c-MET (MET proto-oncogene) status [Count of Participants; unit: Participants] — c-MET status was determined by immunohistochemistry (IHC) and fluorescence in situ hybridization (FISH) methods. cMET staining by IHC is scored from 0 (no staining) to 3+ (staining with strong intensity).
  As introduced in Protocol Amendment 2, c-MET positivity (c-MET High) was defined as IHC intensity score 3+ in >=50% of tumor cells or c-MET IHC intensity score 2+ in >=50% of tumor cells only if they have in addition MET gene copy number >=5 as detected by FISH or MET gene copy number >=5 by FISH and unknown c-MET IHC results.
  c-MET Low was defined as not fulfilling c-MET high criteria.
  Participants
    c-MET High | 2 | 8 | 2 | 12
    c-MET Low | 6 | 20 | 0 | 26

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression (TTP) by Investigator Assessment Per RECIST v1.1
Description: TTP is defined as the time from the date of treatment start to the date of the first documented radiological confirmation of disease progression or death due to underlying cancer. Tumor response was based on investigator assessment per Response Evaluation Criteria In Solid Tumors (RECIST) v1.1. For RECIST v1.1, Progressive disease (PD) = At least a 20% increase in the sum of diameters of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. In addition, the sum must also demonstrate an absolute increase of at least 5 mm. If a patient had not had the event at the date of analysis cut-off or when he/she received any further anti-neoplastic therapy, TTP was censored at the time of the last adequate assessment. TTP was estimated using the Kaplan-Meier method.
Time Frame: Up to approximately 8 years and 2 months
Population: All patients who received at least one dose of INC280. Patients were analyzed according to the treatment group defined in the study protocol to which they were assigned at baseline: Dose-Determining part and Dose Expansion part. In alignment with the primary objective of the study, efficacy was analyzed in the dose expansion part based on the level of c-MET expression, independently of the formulation received, the capsule or the tablet that was introduced later to facilitate the dosing.
Measure: Median (90% Confidence Interval); unit: months
Groups:
- Dose Determining: Patients enrolled in the Dose Determining part of the study
- Dose Expansion: c-MET High: Patients enrolled in the Dose Expansion part of the study with c-MET High
- Dose Expansion: c-MET Low: Patients enrolled in the Dose Expansion part of the study with c-MET Low
- Dose Expansion: All Patients: Patients enrolled in the Dose Expansion part of the study (c-MET High and c-MET Low)
Arm/Group | Dose Determining | Dose Expansion: c-MET High | Dose Expansion: c-MET Low | Dose Expansion: All Patients
Number analyzed (Participants) | 8 | 10 | 20 | 30
months | NA [NA to NA] — Not estimable due to insufficient number of participants with events | 3.6 [2.0 to 7.7] | 2.1 [1.9 to 2.2] | 2.2 [2.0 to 3.2]

2. Secondary Outcome: Overall Response Rate (ORR) by Investigator Assessment Per RECIST 1.1
Description: Tumor response was based on local investigator assessment per RECIST v1.1. ORR per RECIST v1.1 is defined as the percentage of participants with a best overall response (BOR) of Complete Response (CR) or Partial Response (PR).
  For RECIST v1.1, CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to approximately 8 years and 2 months
Population: All patients who received at least one dose of INC280. Patients were analyzed according to the treatment group defined in the protocol to which they were assigned at baseline: Dose-Determining part and Dose Expansion part. In alignment with the secondary efficacy objective of the study, efficacy was analyzed in the dose expansion part based on the level of c-MET expression, independently of the formulation received, the capsule or the tablet that was introduced later to facilitate the dosing.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Dose Determining | Dose Expansion: c-MET High | Dose Expansion: c-MET Low | Dose Expansion: All Patients
Number analyzed (Participants) | 8 | 10 | 20 | 30
Percentage of participants | 0 [0.0 to 36.9] | 30.0 [6.7 to 65.2] | 0 [0.0 to 16.8] | 10.0 [2.1 to 26.5]

3. Secondary Outcome: Disease Control Rate (DCR) by Investigator Assessment Per RECIST 1.1
Description: Tumor response was based on local investigator assessment per RECIST v1.1. DCR is defined as the percentage of participants with a BOR of Complete Response (CR), Partial Response (PR) and Stable Disease (SD).
  For RECIST v1.1, CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters; SD= Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progression).
Time Frame: Up to approximately 8 years and 2 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Dose Determining | Dose Expansion: c-MET High | Dose Expansion: c-MET Low | Dose Expansion: All Patients
Number analyzed (Participants) | 8 | 10 | 20 | 30
Percentage of participants | 25.0 [3.2 to 65.1] | 50.0 [18.7 to 81.3] | 25.0 [8.7 to 49.1] | 33.3 [17.3 to 52.8]

4. Secondary Outcome: Progression-Free Survival (PFS) by Investigator Assessment Per RECIST 1.1
Description: PFS is defined as the time from date of first study treatment intake to the date of the first radiologically documented progression or death due to any cause or initiation of new antineoplastic therapy.
  If a patient did not have an event, PFS was censored at the date of the last adequate tumor assessment.
  PFS was analyzed using Kaplan-Meier estimates.
Time Frame: Up to approximately 8 years and 2 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Determining | Dose Expansion: c-MET High | Dose Expansion: c-MET Low | Dose Expansion: All Patients
Number analyzed (Participants) | 8 | 10 | 20 | 30
months | NA [NA to NA] — Not estimable due to insufficient number of participants with events | 3.6 [1.2 to NA] — Not estimable due to insufficient number of participants with events | 2.1 [0.9 to 3.2] | 2.2 [1.6 to 4.9]

5. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from date of first study treatment intake to date of death due to any cause. If a patient was not known to have died, survival was censored at the date of last contact.
  OS was analyzed using the Kaplan-Meier method.
Time Frame: Up to approximately 8 years and 2 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Determining | Dose Expansion: c-MET High | Dose Expansion: c-MET Low | Dose Expansion: All Patients
Number analyzed (Participants) | 8 | 10 | 20 | 30
months | NA [NA to NA] — Not estimable due to insufficient number of participants with events | 6.3 [2.1 to NA] — Not estimable due to insufficient number of participants with events | 5.8 [3.1 to 8.1] | 5.8 [3.2 to 8.1]

6. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Number of participants with AEs (any AE regardless of seriousness) and SAEs, including changes from baseline in vital signs, electrocardiograms and laboratory results qualifying and reported as AEs.
Time Frame: From first dose of study drug to 30 days after last dose, up to approximately 8 years and 2 months
Population: Safety Set: All patients who received at least one dose of INC280. Patients were analyzed according to the treatment they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | CINC280 300 mg BID Capsule | CINC280 600 mg BID Capsule | CINC280 400 mg BID Tablet
Number analyzed (Participants) | 9 | 27 | 2
Participants
  AEs | 9 | 27 | 2
  Treatment-related AEs | 7 | 17 | 1
  SAEs | 6 | 13 | 1
  Treatment-related SAEs | 1 | 1 | 0
  Fatal SAEs | 1 | 3 | 1

7. Secondary Outcome: Number of Participants With Dose Reductions and Dose Interruptions of CINC280
Description: For patients who did not tolerate the protocol-specified dosing scheme, dose adjustments and interruptions were permitted.
  Number of participants with dose reductions and dose interruptions of CINC280 is reported in this table.
Time Frame: From first dose of study drug to last dose, up to approximately 8 years and 1 month
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | CINC280 300 mg BID Capsule | CINC280 600 mg BID Capsule | CINC280 400 mg BID Tablet
Number analyzed (Participants) | 9 | 27 | 2
Participants
  At least one dose reduction and/or interruption | 6 | 18 | 1
  At least one dose reduction | 1 | 9 | 1
  At least one dose interruption | 6 | 17 | 1

8. Secondary Outcome: Dose Intensity of INC280
Description: Dose intensity of INC280 was calculated as actual cumulative dose in milligrams divided by duration of exposure in days.
Time Frame: From first dose of study drug to last dose, up to approximately 8 years and 1 month
Population: as for outcome 6
Measure: Median (Full Range); unit: mg/day
Arm/Group | CINC280 300 mg BID Capsule | CINC280 600 mg BID Capsule | CINC280 400 mg BID Tablet
Number analyzed (Participants) | 9 | 27 | 2
mg/day | 600.0 [450 to 957] | 1200.0 [721 to 1200] | 674.2 [548 to 800]

9. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of INC280 in the Dose-Determining Part
Description: Pharmacokinetic (PK) parameters were calculated based on INC280 plasma concentrations by using non-compartmental methods. Cmax is defined as the maximum (peak) observed plasma concentration following a dose.
Time Frame: pre-dose, 30 minutes and 1, 2, 4, 6 and 8 hours after morning dose and 12 hours after evening dose on Cycle 1 Day 1 and Cycle 1 Day 15. The duration of one cycle was 21 days.
Population: Patients in the pharmacokinetic analysis set (PAS) with an available value for the outcome measure. PAS consists of all patients who provided an evaluable PK profile. A profile is considered evaluable if all the following conditions are satisfied: patient received at least one dose of the planned treatments, patient provided at least one primary PK parameter and patient did not vomit within 4 hours after the dosing of INC280. Full PK blood samples were not collected in the Dose-Expansion Part
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | CINC280 300 mg BID Capsule
Number analyzed (Participants) | 8
ng/mL
  Cycle 1 Day 1 | 2140 (105.4)
  Cycle 1 Day 15: number analyzed (Participants) | 6
  Cycle 1 Day 15 | 2530 (86.6)

10. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of INC280 in the Dose-Determining Part
Description: PK parameters were calculated based on INC280 plasma concentrations by using non-compartmental methods. Tmax is defined as the time to reach maximum (peak) plasma concentration following a dose. Actual recorded sampling times were considered for the calculations.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Median (Full Range); unit: hours
Arm/Group | CINC280 300 mg BID Capsule
Number analyzed (Participants) | 8
hours
  Cycle 1 Day 1 | 2 [0.5 to 4]
  Cycle 1 Day 15: number analyzed (Participants) | 6
  Cycle 1 Day 15 | 2 [1 to 2.03]

11. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to 12 Hours (AUC0-12h) of INC280 in the Dose-Determining Part
Description: PK parameters were calculated based on INC280 plasma concentrations by using non-compartmental methods. The linear trapezoidal method was used for AUC0-12h calculation. A dosing interval was 12 hours for twice daily dosing.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | CINC280 300 mg BID Capsule
Number analyzed (Participants) | 7
hr*ng/mL
  Cycle 1 Day 1 | 7740 (72.2)
  Cycle 1 Day 15: number analyzed (Participants) | 6
  Cycle 1 Day 15 | 12300 (84.8)

12. Secondary Outcome: Apparent Plasma Clearance (CL/F) of INC280 in the Dose-Determining Part
Description: PK parameters were calculated based on INC280 plasma concentrations by using non-compartmental methods. Apparent drug clearance from the plasma was calculated as dose/AUCinf.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mL/hr
Arm/Group | CINC280 300 mg BID Capsule
Number analyzed (Participants) | 7
mL/hr
  Cycle 1 Day 1 | 46000 (38100)
  Cycle 1 Day 15: number analyzed (Participants) | 0

13. Secondary Outcome: Terminal Elimination Half-life (T1/2) of INC280 in the Dose-Determining Part
Description: PK parameters were calculated based on INC280 plasma concentrations by using non-compartmental methods. Elimination half-life (T1/2) values were calculated as natural logarithm (ln) 2/terminal elimination rate constant.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | CINC280 300 mg BID Capsule
Number analyzed (Participants) | 7
hours
  Cycle 1 Day 1 | 2.27 (0.437)
  Cycle 1 Day 15: number analyzed (Participants) | 6
  Cycle 1 Day 15 | 4.98 (2.00)

14. Secondary Outcome: Accumulation Ratio (Racc) of INC280 in the Dose-Determining Part
Description: PK parameters were calculated based on INC280 plasma concentrations by using non-compartmental methods. Accumulation ratio of drug exposure was calculated as AUC0-12h on Cycle 1 Day 15 divided by AUC0-12h on Cycle 1 Day 1.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | CINC280 300 mg BID Capsule
Number analyzed (Participants) | 5
ratio | 1.56 (0.275)

15. Post Hoc Outcome: All-Collected Deaths
Description: On-treatment deaths were collected from start of treatment to 30 days after last dose.
  Survival follow-up deaths were collected from day 31 after last dose of study treatment until end of study.
  All deaths refer to the sum of on-treatment deaths plus survival follow-up deaths.
Time Frame: On-treatment: Up to approximately 8 years and 2 months. Survival follow-up: Up to approximately 8 years and 2 months.
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | CINC280 300 mg BID Capsule | CINC280 600 mg BID Capsule | CINC280 400 mg BID Tablet
Number analyzed (Participants) | 9 | 27 | 2
participants
  On-treatment deaths | 1 | 5 | 1
  Survival follow-up deaths: number analyzed (Participants) | 8 | 22 | 1
  Survival follow-up deaths | 8 | 17 | 1
  All deaths | 9 | 22 | 2

ADVERSE EVENTS:
Time Frame: Adverse events and deaths in the on-treatment period were collected from first dose of study treatment to 30 days after last dose, up to approximately 8 years and 2 months. Deaths were collected in the survival follow-up from day 31 after last dose of study treatment until the end of the study, up to approximately 8 years and 2 months. These are not considered AEs.
Description: Patients were analyzed according to the treatment they actually received (Safety Set).
  Deaths in the survival follow-up are not considered Adverse Events.
Groups:
- CINC280 300 mg BID Capsule - On-treatment; CINC280 600 mg BID Capsule - On-treatment; CINC280 400 mg BID Tablet - On-treatment: AEs collected during on-treatment period (up to 30 days after last dose).
- CINC280 300 mg BID Capsule - Survival Follow-up; CINC280 600 mg BID Capsule - Survival Follow-up; CINC280 400 mg BID Tablet - Survival Follow-up: Deaths collected in the survival follow-up period (starting from day 31 after last dose). No AEs were collected during this period.
Arm/Group | CINC280 300 mg BID Capsule - On-treatment | CINC280 600 mg BID Capsule - On-treatment | CINC280 400 mg BID Tablet - On-treatment | CINC280 300 mg BID Capsule - Survival Follow-up | CINC280 600 mg BID Capsule - Survival Follow-up | CINC280 400 mg BID Tablet - Survival Follow-up
All-Cause Mortality (participants affected / at risk) | 1/9 | 5/27 | 1/2 | 8/8 | 17/22 | 1/1
Serious Adverse Events (participants affected / at risk) | 6/9 | 13/27 | 1/2 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 9/9 | 27/27 | 2/2 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CINC280 300 mg BID Capsule - On-treatment (N=9) | CINC280 600 mg BID Capsule - On-treatment (N=27) | CINC280 400 mg BID Tablet - On-treatment (N=2) | CINC280 300 mg BID Capsule - Survival Follow-up (N=0) | CINC280 600 mg BID Capsule - Survival Follow-up (N=0) | CINC280 400 mg BID Tablet - Survival Follow-up (N=0)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | NA | NA | NA
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | NA | NA | NA
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | NA | NA | NA
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | NA | NA | NA
Varices oesophageal (Gastrointestinal disorders) | 1 | 1 | 0 | NA | NA | NA
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
General physical health deterioration (General disorders) | 0 | 0 | 1 | NA | NA | NA
Bile duct stenosis (Hepatobiliary disorders) | 0 | 1 | 0 | NA | NA | NA
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0 | NA | NA | NA
Hepatic haemorrhage (Hepatobiliary disorders) | 1 | 0 | 0 | NA | NA | NA
Hepatic mass (Hepatobiliary disorders) | 0 | 1 | 0 | NA | NA | NA
Biliary tract infection (Infections and infestations) | 0 | 1 | 0 | NA | NA | NA
Pneumonia (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Sepsis (Infections and infestations) | 0 | 1 | 0 | NA | NA | NA
Septic shock (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Blood creatinine increased (Investigations) | 0 | 1 | 0 | NA | NA | NA
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | NA | NA | NA
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | NA | NA | NA
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | NA | NA | NA
Headache (Nervous system disorders) | 0 | 0 | 1 | NA | NA | NA
Spinal cord compression (Nervous system disorders) | 0 | 1 | 0 | NA | NA | NA
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 0 | NA | NA | NA
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0 | NA | NA | NA
Hypovolaemic shock (Vascular disorders) | 1 | 0 | 0 | NA | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CINC280 300 mg BID Capsule - On-treatment (N=9) | CINC280 600 mg BID Capsule - On-treatment (N=27) | CINC280 400 mg BID Tablet - On-treatment (N=2) | CINC280 300 mg BID Capsule - Survival Follow-up (N=0) | CINC280 600 mg BID Capsule - Survival Follow-up (N=0) | CINC280 400 mg BID Tablet - Survival Follow-up (N=0)
Anaemia (Blood and lymphatic system disorders) | 3 | 6 | 0 | NA | NA | NA
Leukopenia (Blood and lymphatic system disorders) | 0 | 4 | 0 | NA | NA | NA
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | NA | NA | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 3 | 0 | NA | NA | NA
Visual field defect (Eye disorders) | 0 | 0 | 1 | NA | NA | NA
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 0 | NA | NA | NA
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0 | NA | NA | NA
Ascites (Gastrointestinal disorders) | 1 | 4 | 0 | NA | NA | NA
Constipation (Gastrointestinal disorders) | 2 | 6 | 1 | NA | NA | NA
Diarrhoea (Gastrointestinal disorders) | 5 | 8 | 0 | NA | NA | NA
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Lip dry (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Nausea (Gastrointestinal disorders) | 6 | 9 | 1 | NA | NA | NA
Peptic ulcer (Gastrointestinal disorders) | 0 | 2 | 0 | NA | NA | NA
Vomiting (Gastrointestinal disorders) | 4 | 9 | 1 | NA | NA | NA
Fatigue (General disorders) | 3 | 6 | 1 | NA | NA | NA
Oedema peripheral (General disorders) | 2 | 4 | 0 | NA | NA | NA
Peripheral swelling (General disorders) | 0 | 3 | 0 | NA | NA | NA
Pyrexia (General disorders) | 1 | 5 | 0 | NA | NA | NA
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 4 | 0 | NA | NA | NA
Bronchitis (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | NA | NA | NA
Alanine aminotransferase increased (Investigations) | 0 | 7 | 1 | NA | NA | NA
Amylase increased (Investigations) | 0 | 3 | 0 | NA | NA | NA
Aspartate aminotransferase increased (Investigations) | 1 | 12 | 0 | NA | NA | NA
Bilirubin conjugated increased (Investigations) | 0 | 2 | 0 | NA | NA | NA
Blood albumin decreased (Investigations) | 0 | 2 | 0 | NA | NA | NA
Blood bilirubin increased (Investigations) | 2 | 7 | 0 | NA | NA | NA
Blood cholesterol increased (Investigations) | 1 | 0 | 0 | NA | NA | NA
Blood creatinine increased (Investigations) | 3 | 7 | 0 | NA | NA | NA
Hepatitis B DNA increased (Investigations) | 0 | 2 | 0 | NA | NA | NA
Lipase increased (Investigations) | 0 | 2 | 0 | NA | NA | NA
Neutrophil count decreased (Investigations) | 0 | 2 | 0 | NA | NA | NA
Platelet count decreased (Investigations) | 0 | 4 | 0 | NA | NA | NA
Weight decreased (Investigations) | 2 | 2 | 0 | NA | NA | NA
Weight increased (Investigations) | 0 | 2 | 1 | NA | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 3 | 9 | 0 | NA | NA | NA
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0 | NA | NA | NA
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | NA | NA | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | NA | NA | NA
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 7 | 0 | NA | NA | NA
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | NA | NA | NA
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | NA | NA | NA
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | NA | NA | NA
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | NA | NA | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | NA | NA | NA
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | NA | NA | NA
Dizziness (Nervous system disorders) | 0 | 2 | 0 | NA | NA | NA
Headache (Nervous system disorders) | 0 | 0 | 1 | NA | NA | NA
Syncope (Nervous system disorders) | 1 | 0 | 0 | NA | NA | NA
Insomnia (Psychiatric disorders) | 1 | 5 | 1 | NA | NA | NA
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 0 | NA | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | NA | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA | NA | NA
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA | NA | NA
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA | NA | NA
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | NA | NA | NA
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | NA | NA | NA
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | NA | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. Novartis does not prohibit any investigator from publishing. Any publications from a single site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-05-16): https://cdn.clinicaltrials.gov/large-docs/27/NCT01737827/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-28): https://cdn.clinicaltrials.gov/large-docs/27/NCT01737827/SAP_001.pdf